CLINICAL TRIAL: NCT02701647
Title: Repetitive Transcranial Magnetic Stimulation Promotes Gait Training in People With Parkinson's Disease - a Randomised Controlled Trial
Brief Title: Effects of Combined rTMS and Treadmill Training in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20140423002
Record Dates: First submitted 2016-01-19; First posted 2016-03-08 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2018-06

CONDITIONS: Parkinson's Disease
Keywords: Transcranial Magnetic Stimulation; metaplasticity; gait training
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25Hz-TT (Experimental): Participants will receive 4s train of 25-Hz rTMS pulses with 50s inter-train interval, with an intensity of 80% resting motor threshold (RMT). Participant will receive a total of 600 rTMS pulses in 6 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS); Other: Treadmill training
- 1Hz-TT (Experimental): Participants will receive a total of 600 1-Hz rTMS pulses in 10 minutes for each hemisphere and a total of 1200 pulses ,with an intensity of 80% RMT, followed by 30 minutes of treadmill training.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS); Other: Treadmill training
- Sham-TT (Sham Comparator): Sham rTMS will be applied over the same site as for real rTMS, however, with the cable of the coil disconnected. Another figure-of-eight coil using the same stimulation parameters (intensity, time, and frequency) as per 25Hz-TT group will be placed posterior to the subject's neck with the handle pointing backward to produce the same clicking sound effect. Sham rTMS will be followed by 30 minutes of treadmill training.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS); Other: Treadmill training

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Repetitive TMS (rTMS) is a painless and non-invasive technique for activation of cerebral cortex based on the principle of electromagnetic induction of an electric field in the brain. rTMS will be delivered to the scalp over the leg area of the bilateral motor cortex by using a Magstim Rapid magnetic stimulator. (Magstim Company, Whitland, UK) and 90 mm double cone coil.
Other: Treadmill training — Participants will proceed to 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. 80% of participant's over ground maximum walking speed will be halved and used for warm-up. After warming up, walking speed will be increased by 0.2 km/h every 5 minutes. Progression will be given if patients could tolerate the belt speed with appropriate step length and walk with good stability for 5 minutes. Participants will maintain the maximum speed achieved for the rest of the session or adjusted as needed. Positive verbal feedback will be given to encourage large strides and upright posture during training. The participants will be instructed to walk on treadmill without holding onto the handrails if possible. Participants will perform warm up and cool down exercise to minimize training related-injury.

SUMMARY:
The purpose of this study is to investigate whether the beneficial effect of treadmill training on people with Parkinson's disease can be enhanced by high- and low-frequency repetitive transcranial magnetic stimulation (rTMS).

DETAILED DESCRIPTION:
This is a randomised placebo-controlled trial. Fifty-one participants with Parkinson's disease (PD) will be recruited from the Hong Kong PD association, a self-help group and movement disorders clinic of 3 local hospitals. Written informed consent in accordance with the Declaration of Helsinki will be obtained from all participants. Eligible participants will be randomly assigned into one of the three groups: 1Hz-TT, 25Hz-TT, and sham-TT upon recruitment. Randomisation will be generated by a computer program and group assignment will be blinded to both participants and assessor. Participant will receive either 1-Hz, 25-Hz, or sham rTMS which will last for about 20 minutes followed by 30 minutes treadmill walking training for 12 sessions, 4 times per week for 3 weeks. All assessments will be conducted 1 week before intervention and 1 day after completion of intervention, after 1-month training and at 3-month post training.

The sample size calculation is based on the significant findings of the gait speed reported by Yang et al (2013). A two-way repeated measures ANOVA design with between-subject group effect (3 levels) and within-subject time effect (4 levels) determines that 15 subjects per group are required to achieve 85% power to test the interaction effect between groups and time effect with a 5% significance level and the effect size is 0.2. By assuming 10% dropout rate, 17 subjects will be required per group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease by a neurologist
* had been stable on anti-Parkinsonian medication
* able to walk independently for 30 meters

Exclusion Criteria:

* severe co-morbidity that may interfere with their ability to participate including significant orthopaedic or rheumatological conditions or disorders of peripheral nervous systems that may interfere with mobility or balance performance
* a diagnosis of neurological disease other than PD
* a history of psychiatric disorders
* the impossibility of inducing motor evoked potentials (MEPs)
* a score of less than 24 on the Mini-Mental State Examination
* contraindication to TMS including personal or family history of seizure disorder, metal in the head, implants of medical devices such as cardiac pacemakers or medical pumps, females subjects who are pregnant, a history of neurosurgery
* subjects with irrepressible tremor and / or dyskinesia

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mak, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Rehabilitation Sciences, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with researcher who provide a methodologically sound proposal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication
Access Criteria: request through email

REFERENCES:
- [Background] Yang YR, Tseng CY, Chiou SY, Liao KK, Cheng SJ, Lai KL, Wang RY. Combination of rTMS and treadmill training modulates corticomotor inhibition and improves walking in Parkinson disease: a randomized trial. Neurorehabil Neural Repair. 2013 Jan;27(1):79-86. doi: 10.1177/1545968312451915. Epub 2012 Jul 10. PMID 22785003

RESULTS

PARTICIPANT FLOW:
Groups:
- 25-Hz rTMS: Participants received 4s train of 25-Hz repetitive Transcranial magnetic stimulation pulses with 50s inter-train intervals. Participant received a total of 600 rTMS pulses in 6 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.Treadmill training: Participants proceeded with 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. Walking speed on treadmill was increased by 0.2km/h every 5 minutes provided that participants could tolerate the belt speed with appropriate step length and walk with good stability. The maximum achieved speed was then maintained for the rest of the session or adjusted as needed.
- 1-Hz rTMS: Participants received a total of 600 1-Hz repetitive Transcranial magnetic stimulation pulses in 10 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.
  Treadmill training: Participants proceeded with 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. Walking speed on treadmill was increased by 0.2km/h every 5 minutes provided that participants could tolerate the belt speed with appropriate step length and walk with good stability. The maximum achieved speed was then maintained for the rest of the session or adjusted as needed.
- Sham rTMS: Sham repetitive Transcranial magnetic stimulation was applied over the same site as for real rTMS , however, with the cables of the coil disconnected. Another figure-of-eight coil using the same stimulation parameters (intensity, time, and frequency) as 25-Hz group was placed posterior to the subject's neck with the handle pointing backward to produce the same clicking sound effect as 25-Hz group. Sham rTMS will be followed by 30 minutes of treadmill training.
  Treadmill training: Participants proceeded with 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. Walking speed on treadmill was increased by 0.2km/h every 5 minutes provided that participants could tolerate the belt speed with appropriate step length and walk with good stability. The maximum achieved speed was then maintained for the rest of the session or adjusted as needed.
Period: Overall Study
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Started | 17 | 17 | 17
Completed | 17 | 17 | 16 (One participant from sham-TT withdraw due a back injury unrelated to study.)
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 25-Hz rTMS: Participants received 4s train of 25-Hz repetitive Transcranial magnetic stimulation pulses with 50s inter-train intervals. Participant received a total of 600 rTMS pulses in 6 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.
  Participants will proceed to 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. 80% of participant's over ground maximum walking speed will be halved and used for warm-up. After warming up, walking speed will be increased by 0.2 km/h every 5 minutes. Progression will be given if patients could tolerate the belt speed with appropriate step length and walk with good stability for 5 minutes. Maximum achieved speed will be maintained followed by 0.5 km/h decrements. Participants will maintain the rest of the treadmill session with this speed or further adjustment will be made if participants are unable to maintain. Positive verbal feedback
- Sham rTMS: Sham repetitive Transcranial magnetic stimulation was applied over the same site as for real rTMS , however, with the cables of the coil disconnected. Another figure-of-eight coil using the same stimulation parameters (intensity, time, and frequency) as 25-Hz group will be placed posterior to the subject's neck with the handle pointing backward to produce the same clicking sound effect as 25-Hz group. Sham rTMS will be followed by 30 minutes of treadmill training.
  Treadmill training: Participants proceeded with 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. Walking speed on treadmill was increased by 0.2km/h every 5 minutes provided that participants could tolerate the belt speed with appropriate step length and walk with good stability. The maximum achieved speed was then maintained for the rest of the session or adjusted as needed.
- Total: Total of all reporting groups
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS | Total
Number analyzed (Participants) | 17 | 17 | 16 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 11 | 35
  >=65 years | 4 | 6 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.8) | 62.1 (5.7) | 62.1 (5.7) | 62.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 24
  Male | 10 | 9 | 7 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 17 | 17 | 16 | 50
Disease duration (no. of years of diagnosis of PD) [Mean (Standard Deviation); unit: years] | 5.2 (3.4) | 7.5 (4.9) | 6.9 (3.3) | 6.5 (4.0)
daily levodopa equivalent dose [Mean (Standard Deviation); unit: mg/day] | 484.2 (336.4) | 512.5 (359.9) | 493.3 (523.9) | 496.8 (404.2)

OUTCOME MEASURES:

1. Primary Outcome: Fastest Walking Speed
Description: Each participant is instructed to walk for 14 meters at their fastest walking speed for three trials. The time taken for the middle 10 meter was recorded. The average of three trials is used for analysis.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention, 3 month post-intervention
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- 25-Hz rTMS: Participants received 4s train of 25-Hz repetitive Transcranial magnetic stimulation pulses with 50s inter-train intervals. Participant received a total of 600 rTMS pulses in 6 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.
- 1-Hz rTMS: Participants received a total of 600 1-Hz repetitive Transcranial magnetic stimulation pulses in 10 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.
- Sham rTMS: Sham repetitive Transcranial magnetic stimulation will was applied over the same site as for real rTMS , however, with the cables of the coil disconnected. Another figure-of-eight coil using the same stimulation parameters (intensity, time, and frequency) as 25-Hz group with another coil placed posterior to the subject's neck with the handle pointing backward to produce the same clicking sound effect. Sham rTMS will be followed by 30 minutes of treadmill training.
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 17 | 16
cm/s
  Baseline | 149.5 (24.7) | 153.1 (27.3) | 156.1 (30.2)
  1 day Post intervention | 164.3 (26.3) | 167.3 (34.0) | 160.7 (33.3)
  1 month post intervention | 167.8 (26.4) | 170.6 (35.6) | 164.6 (32.3)
  3 month post intervention | 163.2 (31.0) | 169.9 (38.7) | 156.7 (28.0)

2. Secondary Outcome: Timed-Up-and-Go Test (iTUG)
Description: Participants are instructed to stand up from a chair and walk for 7 meters walkway and return back to the chair turn around and sit down.
  Time and gait parameters during TUG were captured by the valid and reliable APDM system, which is a wearable gait and balance analysis system.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- 25Hz-TT: Participants will receive 4s train of 25-Hz rTMS pulses with 50s inter-train interval, with an intensity of 80% resting motor threshold (RMT). Participant will receive a total of 600 rTMS pulses in 6 minutes for each hemisphere and a total of 1200 pulses followed by 30 minutes of treadmill training.
  Repetitive transcranial magnetic stimulation (rTMS): Repetitive TMS (rTMS) is a painless and non-invasive technique for activation of cerebral cortex based on the principle of electromagnetic induction of an electric field in the brain. rTMS will be delivered to the scalp over the leg area of the bilateral motor cortex by using a Magstim Rapid magnetic stimulator. (Magstim Company, Whitland, UK) and 90 mm double cone coil.
  Treadmill training: Participants will proceed to 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. After warming up, walking speed will be increased by 0.2 km/h every 5 minutes.
- 1Hz-TT: Participants will receive a total of 600 1-Hz rTMS pulses in 10 minutes for each hemisphere and a total of 1200 pulses ,with an intensity of 80% RMT, followed by 30 minutes of treadmill training.
  Repetitive transcranial magnetic stimulation (rTMS): Repetitive TMS (rTMS) is a painless and non-invasive technique for activation of cerebral cortex based on the principle of electromagnetic induction of an electric field in the brain. rTMS will be delivered to the scalp over the leg area of the bilateral motor cortex by using a Magstim Rapid magnetic stimulator. (Magstim Company, Whitland, UK) and 90 mm double cone coil.
  Treadmill training: Participants will proceed to 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. After warming up, walking speed will be increased by 0.2 km/h every 5 minutes.
- Sham-TT: Sham rTMS will be applied over the same site as for real rTMS discounnted coil. Anothe coil using the same stimulation parameters as per 25Hz-TT group will be placed posterior to the subject's neck produce the same clicking sound effect. Sham rTMS will be followed by 30 minutes of treadmill training.
  Repetitive transcranial magnetic stimulation (rTMS): Repetitive TMS (rTMS) is a painless and non-invasive technique for activation of cerebral cortex based on the principle of electromagnetic induction of an electric field in the brain. rTMS will be delivered to the scalp over the leg area of the bilateral motor cortex by using a Magstim Rapid magnetic stimulator. (Magstim Company, Whitland, UK) and 90 mm double cone coil.
  Treadmill training: Participants will proceed to 30 minute of treadmill training after rTMS. A safety harness without body weight support will be provided. After warming up, walking speed will be increased by 0.2 km/h every 5 minutes.
Arm/Group | 25Hz-TT | 1Hz-TT | Sham-TT
Number analyzed (Participants) | 17 | 17 | 16
seconds
  Baseline | 20.8 (4.0) | 18.3 (2.5) | 19.3 (2.5)
  1 day Post intervention | 18.4 (2.8) | 17.1 (2.7) | 18.0 (2.1)
  1 month post intervention | 17.7 (2.9) | 17.1 (2.3) | 17.9 (1.8)
  3 month post intervention | 17.9 (2.8) | 16.6 (2.3) | 18.4 (2.1)

3. Secondary Outcome: the Motor Section of Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS III)
Description: MDS-UPDRS III is a valid and reliable clinical test, will be used to evaluate severity of motor symptoms of PD. There are total of 27 items including tremor, rigidity, bradykinesia, postural instability and gait performance. Each item scores from 0-4, with 0 indicates no disability and 4 maximum disabled with total score(s) ranges from 0 to 132.
Time Frame: Baseline, I day post-intervention, 1 month post-intervention and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 17 | 16
score on a scale
  Baseline | 27.9 (10.5) | 27.1 (9.6) | 29.7 (10.6)
  1 day Post intervention | 19.9 (8.5) | 22.2 (7.5) | 27.9 (9.0)
  1 month post intervention | 20.8 (8.9) | 22.5 (7.3) | 27.9 (10.1)
  3 month post intervention | 22.5 (10.1) | 21.9 (7.8) | 27.3 (8.0)

4. Secondary Outcome: Walking Distance in a 2 -Minute Walk Test
Description: The 2 minute walk test will be conducted along a 20 m x 2 m hallway. A line is marked at each end of the walkway to indicate where the person is to turn. Participants will be instructed to " walk as far as possible in 2 minutes". They will be given standardised encouragement at 60 and 90 seconds during walk. Distance walked will be recorded to the nearest meter.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | 25Hz-TT | 1Hz-TT | Sham-TT
Number analyzed (Participants) | 17 | 17 | 16
meter
  Baseline | 147.4 (29.8) | 144.7 (31.3) | 148.7 (25.0)
  1 day post intervention | 160.4 (28.0) | 164.9 (29.8) | 157.3 (31.7)
  1 month post intervention | 166.3 (29.7) | 167.9 (29.7) | 157.9 (29.7)
  3 month post intervention | 163.1 (30.7) | 166.8 (31.2) | 160.5 (28.9)

5. Secondary Outcome: Mini Balance Evaluation Systems Test Scores
Description: Balance performance of participants will be assessed in 4 domains namely anticipatory postural adjustments, postural responses, sensory orientation and gait stability. Each item is rated from 0-2 with a total scores of 28. The Total scores range from 0-28, with higher scores indicate better dynamic balance.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 25Hz-TT | 1Hz-TT | Sham-TT
Number analyzed (Participants) | 17 | 17 | 16
score on a scale
  Baseline | 21.5 (3.4) | 21.8 (2.7) | 21.7 (2.8)
  1 day post intervention | 24.2 (2.5) | 23.8 (2.7) | 22.4 (2.2)
  1 month post intervention | 23.8 (2.8) | 23.5 (2.5) | 22.8 (2.5)
  3 month post intervention | 23.4 (3.0) | 24.1 (2.6) | 23.0 (2.4)

6. Secondary Outcome: Dual-task Timed-Up-and-Go Test (DT-TUG)
Description: For DT-TUG, participants were instructured to repeat the TUG procedure while performing a serial three substraction. Time taken to complete DT-TUG and accuracy of digital counting was recorded. One practice trial was given prior to both TUG and DT-TUG testing and average performance of three trials was used for analysis.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention, 3 month-post intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 17 | 16
seconds
  Baseline | 27.9 (8.8) | 24.0 (7.0) | 25.5 (5.6)
  1 day Post intervention | 23.1 (5.6) | 21.1 (5.2) | 23.4 (4.0)
  1 month post intervention | 21.8 (6.0) | 20.6 (4.7) | 23.9 (3.9)
  3 month post intervention | 22.3 (6.0) | 20.3 (4.6) | 23.9 (3.9)

7. Other Pre Specified Outcome: Cortical Silent Period
Description: Ten suprathreshold TMS stimuli (i.e. 130% RMT) will be delivered while participant performing a 20% isometric maximal contraction of Tibialis Anterior of the more affected side. Cortical silent period (CSP) measures the duration of interruption of electromyography (EMG) activity in the contracting muscle produced by TMS. CSP duration will be determined as the period between the onset of MEP and the return of baseline EMG activity measured 50 ms before the TMS stimulus.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention and 3 months post-intervention
Population: 1 discarded data due to poor quality of data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 17 | 15
milliseconds
  Baseline | 176.5 (50.0) | 164.6 (39.8) | 183.9 (38.9)
  1 day Post intervention | 194.4 (53.2) | 180.6 (39.1) | 175.1 (46.6)
  1 month post intervention | 190.1 (54.5) | 160.1 (41.1) | 189.2 (37.6)
  3 month post intervention | 175.9 (43.2) | 154.6 (46.0) | 182.9 (35.0)

8. Other Pre Specified Outcome: Gradient of the Recruitment Curve ( Also Known as Stimulus-response Curve)
Description: TMS stimuli will be applied at 10% steps between 100% to 160% RMT. 10 stimuli will be delivered at each intensity. Peak to peak amplitude of 10 motor-evoked potentials (MEPs) at each stimulus intensity will be averaged offline.The cut-off intensity is set at 75% of maximum stimulator output due to discomfort perceived by majority of the participants. MEPs will be normalised with the maximal muscle action potential (MMax), which is determined by supramaximal electrical stimulation of the fibular nerve. A scatter graph will be generated with the average amplitude of MEPs as a function of stimulation intensity. The linear trend will be added to generate the linear recruitment curve slope.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention and 3 months post-intervention
Population: 2 sets of discarded data due to poor quality
Measure: Mean (Standard Deviation); unit: millivolts / % maximum stimulator output
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 16 | 15
millivolts / % maximum stimulator output
  Baseline | 0.51 (0.30) | 0.53 (0.39) | 0.61 (0.32)
  1 day Post intervention | 0.58 (0.36) | 0.64 (0.37) | 0.52 (0.40)
  1 month post intervention | 0.70 (0.57) | 0.63 (0.30) | 0.59 (0.43)
  3 month post intervention | 0.74 (0.47) | 0.70 (0.41) | 0.58 (0.45)

9. Other Pre Specified Outcome: Short-interval-intracortical Inhibition
Description: Short-interval-intracortical inhibition (SICI) is another measure of cortical inhibition. In a paired- pulse TMS paradigm, a test pulse will be adjusted to produce MEP of at least 0.5 millivolts which will be delivered preceded by a brief conditioned pulse set at a lower intensity of 80% RMT with inter-stimulus interval of 2 milliseconds. Two stimulators connected via a Bistim module ( Magstim Co.,Whitland, UK) will be used in this test. Ten conditioned MEPs and unconditioned MEPs will be obtained in a random order and were averaged for each condition. SICI is expressed as percentage of unconditioned test MEP amplitude.
Time Frame: Baseline, 1 day post-intervention, 1 month post-intervention and 3 months post-intervention
Population: unable to perform procedure due to small MEPS values for 5 participants
Measure: Mean (Standard Deviation); unit: percentage of Unconditioned MEPs
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
Number analyzed (Participants) | 15 | 14 | 11
percentage of Unconditioned MEPs
  Baseline | 56.4 (27.0) | 49.4 (24.1) | 62.2 (33.1)
  1 day Post intervention | 44.4 (23.0) | 51.4 (28.2) | 76.5 (49.8)
  1 month post intervention | 42.0 (26.9) | 62.6 (31.7) | 89.8 (62.9)
  3 month post intervention | 50.8 (22.8) | 60.7 (39.2) | 74.3 (30.2)

ADVERSE EVENTS:
Time Frame: during intervention, at 1 day post-intervention,1 month post-intervention and at 3 month post-intervention
Arm/Group | 25-Hz rTMS | 1-Hz rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT02701647/Prot_SAP_000.pdf